CLINICAL TRIAL: NCT03898882
Title: The Pharmacokinetics of Oxytocin in Pregnant Women Undergoing Cesarean Delivery - a Feasibility Pilot Study
Brief Title: Pharmacokinetics of Oxytocin at Cesarean Delivery
Acronym: Peacocks
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201810134
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- BMI 20 - 29.9 kg/m2
  Interventions: Drug: oxytocin; Device: Shore durometer
- BMI > 30 kg/m2
  Interventions: Drug: oxytocin; Device: Shore durometer

INTERVENTIONS:
Drug: oxytocin — PK measurements of oxytocin
Device: Shore durometer — The investigators will take serial readings from a digital durometer at the uterine fundus at 3, 6, 9 and 12 minutes following OXT administration to provide data that will inform an estimate of the timing of peak effect. Shore durometers measure the hardness of materials on a scale of 0-100 Shore Units (SU). Preliminary (unpublished) data provided a range of 10-56 SU after oxytocin administration at cesarean delivery. Durometer readings were also shown to correlate positively with the obstetrician's manual assessment of uterine contractility, which is traditionally used to determine the success or failure of uterotonic therapy.

SUMMARY:
The primary objective is to obtain data to inform the design of a population pharmacokinetic study of oxytocin after administration at CD as per standard institutional practice.

DETAILED DESCRIPTION:
In this pilot study the investigators will compare plasma oxytocin concentrations measured in arterial and venous blood, after oxytocin administration at cesarean delivery, in order to assess the validity of venous samples. They will also measure oxytocinase to explore how levels vary around the time of delivery of the placenta and to assess the effect that this may have on the metabolism of oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Term singleton pregnancy
* Age 18-45 years of age
* ASA classification 2 or 3
* Scheduled cesarean delivery under neuraxial anaesthesia

Exclusion Criteria:

* Age or ASA classification outside of inclusion criteria
* Need for general anaesthesia
* Absence of consent
* Inability to communicate in English or other barrier to providing informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be scheduled for cesarean delivery of their baby
Study Population: Pregnant women scheduled for cesarean delivery of their babies at term
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Arterial [OXT] | Scheduled samples during the first 30 minutes after oxytocin administration
  Concentration of oxytocin in arterial samples
Venous [OXT] | Scheduled samples during the first 30 minutes after oxytocin administration
  Concentration of oxytocin in venous samples

SECONDARY OUTCOMES:
Arterial [OXTase] | Scheduled samples during the first 30 minutes after oxytocin administration
  Concentration of oxytocinase in arterial samples
Uterine tone | Scheduled measurements during the first 30 minutes after oxytocin administration
  Uterine tone measured using a Shore Durometer or assessed by obstetrician using numerical rating score (NRS, 0-10)
Hypotension | Measured intraoperatively
  Incidence of systolic BP reduced by 20% from baseline
Nausea & Vomiting | Recorded intraoperatively
  Incidence of nausea and vomiting
EBL | Estimated at the end of surgery
  Estimated blood loss in milliliters

CONTACTS AND LOCATIONS:
Overall Officials: David T Monks, MBChB, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Attilakos G, Psaroudakis D, Ash J, Buchanan R, Winter C, Donald F, Hunt LP, Draycott T. Carbetocin versus oxytocin for the prevention of postpartum haemorrhage following caesarean section: the results of a double-blind randomised trial. BJOG. 2010 Jul;117(8):929-36. doi: 10.1111/j.1471-0528.2010.02585.x. Epub 2010 May 19. PMID 20482535
- [Background] Chiou WL. The phenomenon and rationale of marked dependence of drug concentration on blood sampling site. Implications in pharmacokinetics, pharmacodynamics, toxicology and therapeutics (Part II). Clin Pharmacokinet. 1989 Oct;17(4):275-90. doi: 10.2165/00003088-198917040-00005. No abstract available. PMID 2686884
- [Background] Chiou WL. The phenomenon and rationale of marked dependence of drug concentration on blood sampling site. Implications in pharmacokinetics, pharmacodynamics, toxicology and therapeutics (Part I). Clin Pharmacokinet. 1989 Sep;17(3):175-99. doi: 10.2165/00003088-198917030-00004. PMID 2680213